CLINICAL TRIAL: NCT03648437
Title: Paracetamol And Ibuprofen/Indomethacin in Closing Patent Ductus Arteriosus of Preterm Infants - Randomised, Placebo-controlled Multicentre Trial
Brief Title: Paracetamol And Ibuprofen/Indomethacin in Closing Patent Ductus Arteriosus
Acronym: PAI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The PDA patients have vanished. The last recruitment took place in 2022. In the joint discussion of the principal researchers, it was concluded that PDA patients no longer have to be treated in Finland and the study was terminated.
Sponsor: University of Oulu (Other)
Collaborators: Helsinki University Central Hospital (Other); Turku University Hospital (Other Government); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Outi Aikio, MD, PhD, Docent, Specialist in Peditrics and Neonatology, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 38/2018
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Patent Ductus Arteriosus
Keywords: acetaminophen; ibuprofen; preterm infant; near infra-red spectroscopy; indomethacin
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth | interventions — Acetaminophen; Sodium Chloride; Ibuprofen; Indomethacin; Injections

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, placebo-controlled, double-blind, clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo, 0.45 % saline, is similar to paracetamol, both being clear liquids, so the staff will remain unaware which drug the patient receives. The study drug will be kept and prepared away from the neonatal intensive care unit, at the separate ward 55 office, in a locked cabinet. The study drug will be prepared by the research nurse, the pharmacist of the ward, or during nighttime, by a nurse who does not participate in the study patients' treatment in any way.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pedea 5mg/mL and Paracetamol 10mg/mL (Experimental): Intravenous (IV) ibuprofen 5mg/mL q 24h for 3 days, dosages: 10mg/kg + 5mg/kg + 5mg/kg and IV paracetamol 10mg/mL for 3 days: loading dose 20mg/kg, following 7.5mg/kg q 6h (up to12 doses)
  Interventions: Drug: Paracetamol 10Mg/mL; Drug: Ibuprofen
- Pedea 5mg/mL and 0.45 sodium chloride (Placebo Comparator): IV ibuprofen 5mg/mL q 24h for 3 days, dosages: 10mg/kg + 5mg/kg + 5mg/kg and NaCl 0.45% for 3 days, the same amount in mL as would have been given IV paracetamol
  Interventions: Drug: 0.45% Sodium Chloride; Drug: Ibuprofen
- Indomethacin 25mg/mL and Paracetamol10mg/mL (Experimental): Intravenous (IV) indometahcin 25mg/mL q 24h for 3 days, dosages: 0.2mg/kg + 0.1mg/kg + 0.1mg/kg and IV paracetamol 10mg/mL for 3 days: loading dose 20mg/kg, following 7.5mg/kg q 6h (up to12 doses)
  Interventions: Drug: Paracetamol 10Mg/mL; Drug: Indomethacin
- Indomethacin 25mg/mL and 0.45 sodium chloride (Placebo Comparator): Intravenous (IV) indomethacin 25mg/mL q 24h for 3 days, dosages: 0.2mg/kg + 0.1mg/kg + 0.1mg/kg and NaCl 0.45% for 3 days, the same amount in mL as would have been given IV paracetamol
  Interventions: Drug: 0.45% Sodium Chloride; Drug: Indomethacin

INTERVENTIONS:
Drug: Paracetamol 10Mg/mL — Experimental drug
  Other Names: Paracetamol Fresenius Kabi 10mg/mL infusion solution
  Arms: Indomethacin 25mg/mL and Paracetamol10mg/mL; Pedea 5mg/mL and Paracetamol 10mg/mL
Drug: 0.45% Sodium Chloride — Placebo comparator
  Other Names: NATRIUMKLORID BRAUN 4,5 mg/mL infusion solution
  Arms: Indomethacin 25mg/mL and 0.45 sodium chloride; Pedea 5mg/mL and 0.45 sodium chloride
Drug: Ibuprofen — Standard therapy
  Other Names: Pedea 5mg/mL injection solution
  Arms: Pedea 5mg/mL and 0.45 sodium chloride; Pedea 5mg/mL and Paracetamol 10mg/mL
Drug: Indomethacin — Standard therapy
  Other Names: Liometacen 50mg/2mL injection
  Arms: Indomethacin 25mg/mL and 0.45 sodium chloride; Indomethacin 25mg/mL and Paracetamol10mg/mL

SUMMARY:
The purpose of this pilot trial is to study efficacy and safety of simultaneous intravenous (iv) ibuprofen/indomethacin and paracetamol medications in the closure of patent ductus arteriosus (PDA) in preterm infants. It is randomized, placebo-controlled, double-blind, phase 1, multicenter, clinical trial.

DETAILED DESCRIPTION:
Premature infants (born before 37 weeks gestational age) with patent ductus arteriosus (PDA) are the focus of the study since no trials on the additive efficacy of these two medications on the contraction of ductus arteriosus are available. Preterm infants who are diagnosed to have a hemodynamically significant PDA and who, according to the decision of the attending clinician, need ibuprofen/indomethacin therapy, are eligible to this trial.

If the parents deny the consent, the patient will be treated according to the standard PDA treatment: three days' iv ibuprofen Pedea® 5mg/ml solution infusion (Oulu, Helsinki, Tartu) dosing: 10mg/kg + 5mg/kg + 5mg/kg (q24h); or three days' iv indomethacin (Turku) 0.2mg/kg + 0.1mg/kg + 0.1mg/kg (q24h). In case of any contraindications for ibuprofen/indomethacin, the treatment would be surgical ligation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants (born before 37+0 gestation weeks) who are diagnosed to have a hemodynamically significant PDA and who, according to the decision of the attending clinician, need ibuprofen therapy, are eligible to this trial.

Exclusion Criteria:

* severe malformation or suspected chromosomal defect
* other very severe life-threatening disease (e.g. very severe birth asphyxia or persistent pulmonary hypertension, etc.)

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Ductal closure | Neonatal internsive care unit (NICU) stay up to 12 weeks
  Number of patients with ductal contraction without need for other PDA therapies

SECONDARY OUTCOMES:
Need for ductal therapies | NICU stay up to 12 weeks
  Given ductal therapies after the study drug
Cardiac ultrasound findings | NICU stay up to 12 weeks
  Ductal caliber (mm, mm/kg), LA/Ao ratio
Duration of any ventilation assist | NICU stay up to 12 weeks
  The ventilation assist time pediod
Paracetamol serum levels | Study drug period up to 4 days
  Measured paracetamol concentrations (mg/mL)
Paracetamol side effects | Study drug period plus 7 days, up to 10 days
  Observed adverse events linked to study drug
Long term complications of prematurity | Hospital stay up to 18 weeks
  Moderate-to-severe bronchopulmonary dysplasia, intraventricular hemorrhage grade 2-4, moderate to severe necrotizing enterocolitis, retinopathy of prematurity needing therapy
Other long-term morbidity, and mortality | Hospital stay up to 18 weeks
  Other severe diseases

CONTACTS AND LOCATIONS:
Overall Officials: Outi Aikio, MD, PhD, Principal Investigator — Oulu Univerisity Hospital
Locations (4):
- Finland (4):
  - Helsinki Univeristy Central Hospital, Helsinki
  - Department of Pediatrics, Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harkin P, Harma A, Aikio O, Valkama M, Leskinen M, Saarela T, Hallman M. Paracetamol Accelerates Closure of the Ductus Arteriosus after Premature Birth: A Randomized Trial. J Pediatr. 2016 Oct;177:72-77.e2. doi: 10.1016/j.jpeds.2016.04.066. Epub 2016 May 20. PMID 27215779
- [Background] Juujarvi S, Saarela T, Hallman M, Aikio O. Intravenous paracetamol was associated with closure of the ductus arteriosus in extremely premature infants. Acta Paediatr. 2018 Apr;107(4):605-610. doi: 10.1111/apa.14137. Epub 2017 Nov 17. PMID 29105147
- [Background] Harma A, Aikio O, Hallman M, Saarela T. Intravenous Paracetamol Decreases Requirements of Morphine in Very Preterm Infants. J Pediatr. 2016 Jan;168:36-40. doi: 10.1016/j.jpeds.2015.08.003. Epub 2015 Aug 29. PMID 26323200
- [Background] Aikio O, Harkin P, Saarela T, Hallman M. Early paracetamol treatment associated with lowered risk of persistent ductus arteriosus in very preterm infants. J Matern Fetal Neonatal Med. 2014 Aug;27(12):1252-6. doi: 10.3109/14767058.2013.854327. Epub 2013 Oct 31. PMID 24111688
- [Background] Juujarvi S, Kallankari H, Patsi P, Leskinen M, Saarela T, Hallman M, Aikio O. Follow-up study of the early, randomised paracetamol trial to preterm infants, found no adverse reactions at the two-years corrected age. Acta Paediatr. 2019 Mar;108(3):452-458. doi: 10.1111/apa.14614. Epub 2018 Nov 12. PMID 30325529
- See also: Thesis, Sanna Juujärvi, MB — http://jultika.oulu.fi/Record/isbn978-952-62-2524-1
- See also: Thesis, Pia Härkin, MD — http://jultika.oulu.fi/Record/isbn978-952-62-2025-3

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT03648437/Prot_SAP_001.pdf